CLINICAL TRIAL: NCT02694302
Title: A Multi-center, Parallel and Randomized Design Clinical Trial of Robot-assisted-gait-training (RAGT) in Stroke Patients to Evaluate Its Efficacy, Safety and Superiority Over Conventional Gait Training
Brief Title: Clinical Trial of Robot-assisted-gait-training (RAGT) in Stroke Patients
Acronym: Walkbot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: P&S Mechanics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UMT2013-PS-WB-01
Record Dates: First submitted 2016-02-18; First posted 2016-02-29 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Stroke
Keywords: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Walkbot (Experimental): Walkbot(robot assisted gait training) 30 minutes and conventional physical therapy 30 minutes each per day to be administered 5 times a week for 3 weeks.
  Interventions: Device: Walkbot; Device: Conventional physical therapy
- Conventional physical therapy (Active Comparator): Conventional physical therapy 30 minutes to be administered twice a day, 5 times a week for 3 weeks.
  Interventions: Device: Conventional physical therapy

INTERVENTIONS:
Device: Walkbot — Walkbot(robot assisted gait training) 30 minutes and conventional physical therapy 30 minutes each per day to be administered 5 times a week for 3 weeks.
  Arms: Walkbot
Device: Conventional physical therapy — Conventional physical therapy 30 minutes to be administered twice a day, 5 times a week for 3 weeks.

SUMMARY:
A clinical trial of robot-assisted-gait-training (RAGT) in stroke patients to evaluate its efficacy, safety over conventional gait training.

DETAILED DESCRIPTION:
Robot-assisted-gait-training (RAGT) in stroke patients to evaluate its efficacy, safety over conventional gait training.

Experimental group receives robot-assisted-gait-training and conventional gait training.

Active comparator group receives conventional gait training only as the same number as the experimental group.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 19 and under 80
* Weight under 100kg
* Height less than 200cm
* Able to walk independently before onset of stroke
* Ischemic or hemorrhagic stroke patients
* Patients with motor paralysis and gait disturbance after stroke and seeking rehabilitation treatment
* FAC(Functional Ambulation Category) under 3 (0~2)
* Subacute stroke patients after 3 days and before 3 months of onset
* Be informed of the nature of the study and agreed on written consent voluntarily
* Patients taking medications or scheduled medications due to stroke

Exclusion Criteria:

* Patients with contraindications to weight bearing such as fractures, etc.
* Uncontrolled stage 2 hypertension (systolic over 160 mmHg or diastolic more than 100mmHg) or with uncontrolled orthostatic hypotension
* Patients with cardiopulmonary disease or other underlying diseases that can not tolerate gait training
* Patients with severe skin damage and bedsore on wearing part of the trial device
* Pregnant or breast-feeding
* Participation within 30 days of the other clinical trials
* Patients whom the investigator considers inappropriate to participate in the study

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2014-03; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Functional Ambulation Category(FAC) | 9 weeks from baseline

SECONDARY OUTCOMES:
Motricity Index(MI) | 9 weeks from baseline
10 Meter Walk Test(10MWT) | 9 weeks from baseline
6 Minute Walk Test(6MWT) | 9 weeks from baseline
Medical Research Council(MRC) Scale | 9 weeks from baseline
Modified Ashworth Scale (MAS) | 9 weeks from baseline
Fugl-Meyer Assessment(FMA) of Motor Recovery after Stroke | 9 weeks from baseline
Modified Barthel Index(MBI) | 9 weeks from baseline
National Institutes of Health Stroke Scale (NIHSS) | 9 weeks from baseline
Beck's Depression Inventory test (BDI) | 9 weeks from baseline
Treatment Satisfaction Survey | 9 weeks from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jung Hwan Kim, MD, PhD, Principal Investigator — National Rehabilitation Center, Korea
Locations (2):
- South Korea (2):
  - National Rehabilitation Center, Seoul
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No